CLINICAL TRIAL: NCT02886598
Title: Post-Marketing Surveillance to Evaluate the Safety and Efficacy of Firmagon® (Degarelix) for Injection
Brief Title: Safety and Efficacy of Firmagon® (Degarelix) for Injection
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000260
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Firmagon®: Treatment according to standard clinical practice.
  Interventions: Drug: degarelix

INTERVENTIONS:
Drug: degarelix
  Other Names: Firmagon®

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Firmagon® (degarelix) for injection under the conditions of general clinical practice in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for the treatment of Firmagon® (degarelix) for injection according to the approved product label, and Firmagon® (degarelix) treatment decided before study enrolment. Moreover, patient should have not previously received Firmagon® (degarelix) for injection before the study commencement date at each site. - Indication: treatment of advanced, hormone-dependent prostate cancer.

Exclusion Criteria:

* Patients with previous or concurrent known hypersensitivity to any component of the drug.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who visit department of Urology in hospitals for treatment of prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Gangnam Severance Hospital (there may be other sites in this country), Seoul, South Korea